CLINICAL TRIAL: NCT06399003
Title: A Phase III, Multi-Center, Randomized, Observer-Blind, Active Controlled Non-Inferiority Study to Evaluate the Immunogenicity and Safety of SIBP's MMR Vaccine Compared to GSK MMR Vaccine in Children, 9-11 Months of Age
Brief Title: Comparison Study of SIBP's MMR Vaccine Versus GSK MMR Vaccine in Children Aged 9-11 Months
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Collaborators: Victoria Biomedical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SIBP-MMR-02
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Measles-Mumps-Rubella
Keywords: Measles, Mumps and Rubella; Immunogenicity; Safety; 9-11 months of Age
MeSH Terms: conditions — Measles; Mumps; Rubella | interventions — Measles-Mumps-Rubella Vaccine; Yellow Fever Vaccine

STUDY DESIGN:
Intervention Model Description: The enrolled children will be randomized to three groups in the ratio of 1:1:1 receiving different vaccines.
Who Masked: Outcomes Assessor
Masking Description: This study will have an observer-blinded phase for Group 1 and Group 2 followed by an open label phase from Day 43. Group 3 will remain an open label arm throughout the period of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SIBP MMR vaccine group (Experimental): Received a single dose of SIBP MMR vaccine alone at 1st dose on D1 and licensed Yellow Fever (YF) vaccine alone at 2nd dose on D43.
  Interventions: Biological: SIBP MMR Vaccine; Biological: Yellow Fever Vaccine (Stamaril)
- GSK MMR vaccine group (Active Comparator): Received a single dose of GSK MMR vaccine alone at D1.
  Interventions: Biological: GSK MMR Vaccine (PRIORIX)
- Joint vaccination group (Experimental): Received a single dose of SIBP MMR vaccine co-administered with Yellow Fever vaccine on D1.
  Interventions: Biological: SIBP MMR Vaccine; Biological: Yellow Fever Vaccine (Stamaril)

INTERVENTIONS:
Biological: SIBP MMR Vaccine — This is a live attenuated measles, mumps, and rubella combined vaccine (Shanghai MMR) in a freeze-dried powder form, developed and manufactured by Shanghai Institute of Biological Products. A single dose of 0.5 mL, containing not less than 3.0 log CCID50 of both live measles virus and rubella virus and 4.3 log CCID50 of live mumps virus. 0.5ml per dose.
  Arms: Joint vaccination group; SIBP MMR vaccine group
Biological: GSK MMR Vaccine (PRIORIX) — PRIORIX (combined measles, mumps and rubella vaccine, live, attenuated) is a lyophilized mixed preparation of the attenuated Schwarz measles, RIT 4385 mumps (derived from Jeryl Lynn strain) and Wistar RA 27/3 rubella strains of viruses, separately obtained by propagation either in chick embryo tissue cultures (mumps and measles) or MRC5 human diploid cells (rubella). 0.5ml per dose.
  Arms: GSK MMR vaccine group
Biological: Yellow Fever Vaccine (Stamaril) — This is a live, attenuated, lyophilized yellow fever vaccine manufactured by Sanofi Pasteur Europe, Lyon, France. A single dose of 0.5 mL contains with not less than 1000 IU of yellow fever virus 17D-204 strain. 0.5ml per dose.
  Arms: Joint vaccination group; SIBP MMR vaccine group

SUMMARY:
To evaluate the Immunogenicity and Safety of Shanghai Institute of Biological Products Co., Ltd.'s Measles, Mumps and Rubella (MMR) Vaccine Compared to a Licensed and WHO Prequalified GSK MMR Vaccine in Healthy African Children, 9-11 Months of Age.

DETAILED DESCRIPTION:
This study is designed as a phase III, multi-center, randomized, observer blind active controlled non-inferiority study, enrolling 1200 healthy African children between the ages of 9-11 months. The enrolled children will be randomized to three groups in the ratio of 1:1:1 (400 children in each group) receiving a single dose of SIBP MMR vaccine alone at 1st dose on D1 and licensed YF vaccine alone at 2nd dose on D43 (Group 1, MMR1YF2) or a single dose of GSK MMR vaccine alone at D1 (Group 2, GSK MMR1) or a single dose of SIBP MMR vaccine co-administered with YF vaccine on D1 (Group 3, MMR1YF1). This study will have an observer-blinded phase for Group 1 and Group 2 followed by an open label phase from Day 43. Group 3 will remain an open label arm throughout the period of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female child as established by medical history and clinical examination at enrollment.
* Age: 9-11 months (inclusive) at the time of enrollment
* Parent's/legally acceptable representative's (LAR) ability to read and willingness to provide written informed consent as per the ethical and regulatory requirements of the site.
* Parent confirms intention to stay in the study area for the study duration, bring their child in for the required study visits or to accept a home visit by the study staff.

Exclusion Criteria:

* Presence of fever (defined as axillary temperature ≥ 37.5°C) (temporary exclusion until recovery)
* Acute disease of moderate to severe intensity at the time of enrollment (temporary exclusion until recovery)
* Use of antipyretics within the last 72 hours prior to enrolment (temporary exclusion until recovery)
* Prior (within 6 months) or concurrent participation in another interventional clinical trial during the study
* Presence of severe malnutrition (weight-for-height z-score < -3SD median)
* Positive test for any of the following: HIV, hepatitis B, hepatitis C and syphilis
* Presence of any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological (including severe anemia), endocrine, immunological, dermatological, neurological, cancer, or autoimmune disease) as determined by medical history and / or physical examination which would compromise the participant's health or is likely to result in nonconformance to the protocol.
* Known or suspected impairment of immunological function based on medical history and physical examination.
* Prior receipt or intent to receive measles, mumps, rubella, or yellow fever-containing vaccine during the study vaccination and follow up period up to Day 85 outside the study center.
* Receipt of any vaccine (except OPV and inactivated influenza) within 4 weeks of the day of study vaccination or intent to receive any within 6 weeks after study vaccination.
* Receipt of immunoglobulin therapy and / or blood products in the past 9 months or planned administration during the study period
* Receipt of any immune-modifying or immunosuppressant drugs prior to the first study vaccine dose or planned use during the study. A chronic oral or parenteral use (defined as more than 14 days) of high dose corticosteroids (defined as ≥2 mg/kg of body weight or ≥20 mg/day of prednisone or equivalent for persons who weigh >10 kg) will be exclusionary for the study. Children on inhaled or topical steroids may be permitted to participate in the study.
* Evidence of a clinically significant major congenital anomaly or genetic defect as judged by the investigator.
* Any known or suspected bleeding disorder in the participant that would pose a risk to venipuncture or intramuscular injection.
* History of any neurologic disorders including encephalopathy, epilepsy, and other progressive neurological diseases
* A known or suspected sensitivity or allergy to any components of the investigational product including egg, chicken protein and the antibiotic gentamycin.
* History of severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis.
* Any medical condition in the parent/LAR or child which, in the judgment of the Investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parent(s)'/LAR's ability to give informed consent.

Ages: 9 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
Difference of seropositivity rate | 42 days
  An evaluation of seropositivity rate to Measles, Mumps and Rubella viruses of SIBP MMR vaccine versus GSK MMR vaccine when measured 42 days after vaccination in seronegative children at baseline.

SECONDARY OUTCOMES:
The percentage of immediate adverse events (AEs) | 30 minutes
  The percentage of any adverse events in subjects within 30 minutes after each vaccination.
The percentage of solicited local reactogenicity | 7 days
  The percentage of solicited local reactogenicity in subjects through 7 days after each vaccination.
The percentage of solicited systemic reactogenicity | 14 days
  The percentage of solicited systemic reactogenicity in subjects through 14 days after each vaccination.
The percentage of unsolicited AEs | 42 days
  The percentage of unsolicited AEs in subjects through 42 days after each vaccination.
The percentage of serious adverse events (SAEs) | 42 days
  The percentage of SAEs reported up to 42 days and up to 6 months after first vaccination.
Geometric mean titer (GMT) of Yellow Fever | 42 days
  Geometric mean titer (GMT) for anti-yellow fever virus neutralizing antibodies at baseline and 42 days after vaccination.
Geometric mean concentration (GMC) of Measles | 42 days
  Geometric mean concentration (GMC) for anti-measles IgG antibodies at baseline and 42 days after vaccination.
Geometric mean concentration (GMC) of Mumps | 42 days
  Geometric mean concentration (GMC) for anti-mumps IgG antibodies at baseline and 42 days after vaccination.
Geometric mean concentration (GMC) of Rubella | 42 days
  Geometric mean concentration (GMC) for anti-rubella IgG antibodies at baseline and 42 days after vaccination.
Seropositivity rate of Measles | 42 days
  Seropositivity rate for measles antigen as measured by antibody titers at baseline and 42 days after vaccination.
Seropositivity rate of Mumps | 42 days
  Seropositivity rate for mumps antigen as measured by antibody titers at baseline and 42 days after vaccination.
Seropositivity rate of Rubella | 42 days
  Seropositivity rate for rubella antigen as measured by antibody titers at baseline and 42 days after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Otieno, Doctor, Principal Investigator — Victoria Biomedical Research Institute
Locations (1):
- Victoria Biomedical Research Institute(VIBRI), Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No